CLINICAL TRIAL: NCT00183469
Title: Eight-Month Maintenance Treatment of Bipolar Depression With Lamotrigine or Lamotrigine Plus Divalproex Combination
Brief Title: Maintenance Treatment of Bipolar Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Charles L. Bowden, Professor, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P20MH068662 (NIH); 5P20MH068662 (NIH); DSIR 83-ATSO
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Results first posted 2015-04-20 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-04

CONDITIONS: Bipolar Disorder; Depression
Keywords: Lamotrigine; Divalproex; Antidepressant
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — Lamotrigine; lipoarabinomannan; Valproic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- lamotrigine plus divalproex ER (Active Comparator): Participants will take active lamotrigine and active divalproex ER
  Interventions: Drug: Lamotrigine; Drug: Divalproex (DIV) ER
- lamotrigine plus placebo divalproex ER (Placebo Comparator): Participants will take active lamotrigine and placebo
  Interventions: Drug: Lamotrigine; Drug: Placebo

INTERVENTIONS:
Drug: Lamotrigine — If the participant is naive to LAM, LAM will be started at 25 mg every day for the first 2 weeks, then 50 mg per day for the next 2 weeks. The dose of LAM can be increased to 100 mg at week 5 and increased to maximum of 200 mg at week 6 based on symptoms, tolerability, and ratings of the rating scales. If the participant is already taking LAM, the dose will be increased to up to 200 mg using the same guide lines. Upon randomization the participant in the placebo comparator will have their dosage titrated to doubled since the potentiating effect of the Divalproex will no longer exist. It will remain at this dosage until the end of the study with the possibility of one adjustment for side effects.
  Other Names: Lamictal; (LAM)
Drug: Divalproex (DIV) ER — If the participant is naive to DIV and if LAM was initiated before the start of treatment with DIV, DIV can be started at any point of time in the study provided the participant has been on LAM for at least 2 weeks. DIV will be started at 500 mg and titrated by increments of 500 mg every 3 to 4 days until a therapeutic blood level is attained up to 2500 mg.
  Other Names: Depakote ER; valproic Acid
  Arms: lamotrigine plus divalproex ER
Drug: Placebo — During the randomized phase participants randomized to placebo comparator group will discontinue DIV and will start taking the placebo in the same fashion.
  Other Names: PBO
  Arms: lamotrigine plus placebo divalproex ER

SUMMARY:
This study will compare two different antidepressant treatment regimens to determine which is more effective in reducing symptoms of bipolar depression.

DETAILED DESCRIPTION:
Depression is a serious condition that is often difficult to diagnosis and treat. Bipolar disorder-related depression is especially complex because of the presence of mania symptoms. Lamotrigine and divalproex are commonly prescribed medications for depression. However, their effectiveness in treating bipolar depression has not been thoroughly evaluated. Studies have shown that combining lamotrigine with another antidepressant may be more effective in reducing depressive symptoms than lamotrigine alone. This study will provide participants with either lamotrigine alone or in combination with divalproex and will determine which regimen is more effective in reducing symptoms of bipolar depression.

Participants will be randomly assigned to a daily regimen of either lamotrigine and divalproex or lamotrigine and placebo for 8 months. Participants will be assessed at study entry, at two unspecified times during the study, and at the end of the study. During each assessment, participants will undergo a brief interview and complete a questionnaire about their depressive symptoms, any physical manifestations of their depression, and their overall level of functioning in daily activities.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bipolar disorder I or II
* Experiencing symptoms of depression at study entry OR have experienced symptoms of depression within 6 months prior to study entry
* Willing to use acceptable methods of contraception
* Parent or guardian willing to provide informed consent, if applicable

Exclusion Criteria:

* History of liver disease
* History of substance abuse
* Previous treatment with lamotrigine or divalproex
* Lamotrigine or divalproex intolerance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2004-12; Primary Completion 2009-02 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles L. Bowden, MD, Principal Investigator — 210-567-5405

REFERENCES:
- [Result] Bowden CL, Singh V, Weisler R, Thompson P, Chang X, Quinones M, Mintz J. Lamotrigine vs. lamotrigine plus divalproex in randomized, placebo-controlled maintenance treatment for bipolar depression. Acta Psychiatr Scand. 2012 Nov;126(5):342-50. doi: 10.1111/j.1600-0447.2012.01890.x. Epub 2012 Jun 18. PMID 22708645

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from October 2004 to September 2007 took place in Univ of Texas Health Science Center San Antonio and Center for Healthcare services and television advertisements.
Pre-assignment Details: 1st 8 weeks is Open Label phase. Subjects are either in a depressed episode or have been depressed in last 6 mos. In this phase subjects will take lamotrigine and divalproex ER. Those who remained depressed, or developed an episode, during 2 consecutive visits, were terminated at, or by, week 8.
Groups:
- Double-Blind Lamotrigine and Divalproex ER: Double blind randomized participants will take active lamotrigine and active divalproex Er
- Double-Blind Lamotrigine and Placebo Divalproex ER: Double-Blind randomized Participants will take active lamotrigine and placebo divalproex ER
Period: Overall Study
Arm/Group | Double-Blind Lamotrigine and Divalproex ER | Double-Blind Lamotrigine and Placebo Divalproex ER
Started | 41 | 45
Completed | 13 | 16
Not Completed | 28 | 29

BASELINE CHARACTERISTICS:
Groups:
- Lamotrigine Plus Divalproex ER: Enrolled subjects received lamotrigine and divalproex ER
- Total: Total of all reporting groups
Arm/Group | Lamotrigine Plus Divalproex ER | Lamotrigine Plus Placebo Divalproex ER | Total
Number analyzed (Participants) | 41 | 45 | 86
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 45 | 86
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.6 (11.0) | 42.1 (12.7) | 39.9 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 26 | 47
  Male | 20 | 19 | 39
Region of Enrollment [Number; unit: participants]
  United States | 41 | 45 | 86

OUTCOME MEASURES:

1. Primary Outcome: Mania Rating Scale
Description: Severity of the illness and psychopathological features will be measured by the increase in the SADS Mania Rating Scale, with higher scores representing worse mania. The range of this scale is 0-75.
Time Frame: up to 8 months
Population: all randomized subjects
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Double-Blind Lamotrigine and Divalproex ER | Double-Blind Lamotrigine and Placebo Divalproex ER
Number analyzed (Participants) | 41 | 45
units on a scale | 4.54 (.64) | 5.57 (.6)

ADVERSE EVENTS:
Time Frame: 10/19/2004 - 6/12/2008, 3years 8 months
Description: subject reporting and systematic questionnaires
Groups:
- Lamotrigine Plus Active Divalproex ER: randomized participants will take active lamotrigine and active divalproex Er
- Lamotrigine Plus Placebo Divalproex ER: randomized subjects will take active lamotrigine and placebo divalproex ER
Arm/Group | Lamotrigine Plus Active Divalproex ER | Lamotrigine Plus Placebo Divalproex ER
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/45
Other Adverse Events (participants affected / at risk) | 0/41 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes